CLINICAL TRIAL: NCT06500650
Title: The Effect of Vırtual Reality Application on Visual Skills, Perceived Occupational Performance And Satisfaction ın Elderly People With Mild Cognitive Impairment: A Randomised Controlled Trial
Brief Title: The Effect of Vırtual Reality Application ın Elderly People With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Berkan Torpil, PhD, Associate Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/163
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Intervention Group (Experimental): Virtual reality application and person-centered occupational therapy intervention were applied to the virtual reality intervention group. VR intervention was implemented in a 30 m2 virtual reality unit using a PC Microsoft Kinect and a screen (50" flat LED screen TV) located approximately 1.5 meters away. Kinect can monitor the client's movements in the VR environment in real time by displaying them on the screen. In our study, before starting VR interventions, suitable games for intervention were determined by analyzing which skills each game required and which skills it could develop. Before starting the VR intervention, clients were informed about the games and shown how to play them.
  Interventions: Behavioral: Person-centred Occupational Therapy Intervention
- Person-centred Occupational Therapy Intervention Group (Experimental): Person-centered occupational therapy intervention was applied to both groups according to the evaluation results. The basis of the person-centered occupational therapy intervention is the activities and visual skills that the participants stated in the COPM in the first evaluation and in which they had problems. Person-centered occupational therapy intervention consists of 5 stages: (1) person-centered goal setting, (2) creation of the therapy plan, (3) implementation of interventions, (4) evaluation of results, and (5) obtaining feedback.
  Interventions: Behavioral: Person-centred Occupational Therapy Intervention

INTERVENTIONS:
Behavioral: Person-centred Occupational Therapy Intervention — Person-centred Occupational Therapy Intervention

SUMMARY:
This study was conducted to investigate the effect of virtual reality application on visual skills, perceived occupational performance and satisfaction in elderly individuals with mild cognitive impairment. This study was designed according to the CONSORT statement, which provides a standard method for randomised controlled trial (RCT) design. The study was approved by the Local Ethics Committee. Written informed consent was obtained from all participants before the study.

DETAILED DESCRIPTION:
This study is a single-centre randomised controlled trial involving elderly individuals with mild cognitive impairment in Turkey. The research protocol was approved by the local ethics committee prior to the study. All participants gave written informed consent. This study was designed according to the CONSORT statement, which provides a standardised method for randomised controlled trial (RCT) design.

Participants: For the study, 60 elderly individuals with a diagnosis of HBB were evaluated. Fifty individuals who completed the assessment and met the inclusion/exclusion criteria were included in the study. A virtual reality intervention group (n=25) and a person-centred occupational therapy intervention group (n=25) were formed with the online randomisation application available at https://www.randomizer.org/ by randomly numbering from 1 to 50 with simple random sampling method. Two participants from the person-centred occupational therapy intervention group were excluded from the study because they did not regularly participate in the intervention programme. The study was completed with 48 participants.

Data were analysed with Statistical Package for the Social Sciences (SPSS) version 28.0 statistical package programme. The conformity of the data to normal distribution was tested by Shapiro-Wilk test. Independent Intergroup t test was used to compare normally distributed variables in two independent groups, and Mann Whitney U test was used to compare non-normally distributed variables in two independent groups. As descriptive statistics, mean (±) and standard deviation (X ± SD) values were given for numerical variables and number (n) and percentage (%) values were given for categorical variables.

Multivariate analysis of variance (MANOVA) was used to evaluate the effectiveness of the interventions. It was seen that the prerequisites before MANOVA were met. MANOVA is used to test whether groups formed according to one or more factors show a difference in terms of more than one dependent variable. MANOVA is a powerful multivariate statistic used in experimental research. The use of MANOVA is appropriate when there is a relationship between dependent variables. In this study, Box and Leveni tests, which are the test statistics produced by MANOVA to evaluate the differences between groups, were used to analyse the differences between groups. In the statistical analyses, the significance level was accepted as .05.

ELIGIBILITY:
Inclusion Criteria:

* Being between 65-75 years of age
* Receiving a diagnosis of MCI according to DSM-5
* Being able to read and write
* Ability to understand and follow verbal instructions
* Not having auditory, visual and physical problems that may affect rehabilitation practice and communication

Exclusion Criteria:

* Having a chronic disease that may affect cognitive function
* Participation in any rehabilitation programme (physiotherapy, speech therapy, psychotherapy, etc.) during the study period
* Not being able to participate regularly in the intervention programme during the study period

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
Visual Perception Test Independent of Motor Skills-4 | 30 minutes
  The Motor Skill Independent Visual Perception Test-4 (MVPT-4) is a standardised test (α= 0.80, r=0.53) that assesses visual perception skills without requiring motor or verbal responses. The test consists of 45 items and takes approximately 20 minutes. 4- It can be used in 85+ people. MVPT-4 evaluates five categories of visual perception: visual discrimination, spatial relationship, visual memory, shape-ground, visual proximity. The test result is determined by subtracting the total number of 45. The higher the score, the better the visual perception skill is interpreted.
Canadian Occupational Performance Measure(COPM) | 30 minutes
  COPM, which is most frequently used among occupational therapists, is a standardised measurement tool used to determine the individual's activity performance problems and to measure performance satisfaction. In the COPM, which is a semi-structured interview, individuals evaluate their activity preferences with performance and satisfaction scores given by themselves. Individuals are asked about their activity performance problems and concerns about 3 areas including self-care, productivity and leisure time activities. Up to three problems can be identified in each activity area (self-care, productivity, leisure). Performance and satisfaction scores are again determined by the individual between 1 and 10 points. The Turkish adaptation, validity and reliability study of the COPM was conducted by Torpil et al.

SECONDARY OUTCOMES:
Trail Making Test(TMT) | 25 minutes
  In form A; before the test starts, the numbers from 1 to 8 on the sample application form of the test are asked to be drawn in a way to be followed in order. After the trial test, the participants are asked to combine the numbers from 1 to 25 against time and the time is recorded in seconds when the test is completed. The Turkish validation of the TMT-A was performed by Cangöz et al. The ICC values of the test were found to be 0.78 and 0.99, respectively. In form B, the test consists of a series of circles numbered between 1-13 and circles with letters from A to L on a piece of paper. The person is asked to proceed by matching the numbers and letters from number to letter. The time (in seconds) to complete the combination constitutes the score for the test. The ICC values of the test, which was validated in Turkish by Cangöz et al. were found to be 0.73 and 0.93, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Berkan Torpil, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No